CLINICAL TRIAL: NCT07243652
Title: Cluster Randomized Trial of a Moderate vs High Resource Implementation Strategy to Increase As-needed Post-hospitalization Follow-up for Children With Bronchiolitis
Brief Title: I-DECIDE After Bronchiolitis Hospitalization
Acronym: I-DECIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Eric Coon, Professor of Pediatrics, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPS-2024C1-35425
Record Dates: First submitted 2025-09-29; First posted 2025-11-24 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Bronchiolitis Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Resource Implementation Strategy (Active Comparator)
  Interventions: Other: Moderate-Resource Implementation Strategy
- High-Resource Implementation Strategy (Experimental)
  Interventions: Other: High-Resource Implementation Strategy

INTERVENTIONS:
Other: Moderate-Resource Implementation Strategy — The moderate-resource implementation strategy includes educational outreach (including family-facing materials to support follow-up decision making), audit and feedback (review of clinician performance, captured in a structured report), and materials for clinical decision support.
  Arms: Moderate-Resource Implementation Strategy
Other: High-Resource Implementation Strategy — The high-resource implementation strategy includes all of the moderate resource components, plus two forms of external facilitation: small-group facilitation and expert clinical decision support coach-led facilitation. In total, the high-resource implementation strategy includes educational outreach (including family-facing materials to support follow-up decision-making), audit and feedback (review of clinician performance, captured in a structured report), materials for clinical decision support, small-group facilitation and expert clinical decision support coach-led facilitation.
  Arms: High-Resource Implementation Strategy

SUMMARY:
Although automatic follow-up is a nearly universal practice, research has shown that these visits are often unnecessary after hospitalizations caused by bronchiolitis. Despite endorsement by national pediatric authorities, robust evidence, and family enthusiasm for as-needed (PRN) follow-up, it remains substantially underutilized for children hospitalized for bronchiolitis.

The goal of I-DECIDE is to compare the effects of two multi-component implementation strategies, both of which aim to (a) increase PRN follow-up prescribing by hospitalists (physicians who care for hospitalized children) and (b) decrease unnecessary follow-up visit attendance by families.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of bronchiolitis, discharged by a generalist inpatient service from a non-ICU, non-emergency department, non-step down unit

Exclusion Criteria:

* Children with a history of gestational age <28 weeks, chronic lung disease, complex or hemodynamically significant heart disease, immunodeficiency, or neuromuscular disease
* Children being discharged with home oxygen therapy

Ages: 0 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2700 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Adoption | Within 7 days of hospital discharge
  Proportion of participants who are prescribed PRN follow-up

SECONDARY OUTCOMES:
Sustainment | Within 7 days of hospital discharge
  Proportion of participants who attend a follow-up visit

CONTACTS AND LOCATIONS:
Locations (56):
- United States (56):
  - Children's of Alabama, Birmingham, Alabama
  - Phoenix Children's Hospital - Arrowhead Campus, Glendale, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Adventist Health Lodi Memorial, Lodi, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Children's Hospital Orange County (CHOC), Orange, California
  - University of California Davis Children's Hospital, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - OSF Children's Hospital of Illinois, Peoria, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Baystate Children's Hospital, Springfield, Massachusetts
  - Children's Mercy Kansas City, Kansas City, Missouri
  - Cox Medical Center South, Springfield, Missouri
  - Bryan Medical Center - Children's Nebraska Community site, Lincoln, Nebraska
  - Children's Nebraska, Omaha, Nebraska
  - Children's Hospital at Dartmouth-Hitchcock, Manchester, New Hampshire
  - JM Sanzari Children's Hospital, Hackensack Meridian Children's Health, Hackensack, New Jersey
  - CHOP Pediatric Care at Penn Medicine/Princeton Health, Plainsboro, New Jersey
  - Albany Medical Center, Albany, New York
  - Oishei Children's Hospital, Buffalo, New York
  - Hassenfeld Children's Hospital at NYU Langone, New York, New York
  - University of Rochester Golisano Children's Hospital, Rochester, New York
  - Children's Hospital at Montefiore, The Bronx, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - Children's Hospital of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Texas Children's Hospital - North Campus, Austin, Texas
  - Baylor Scott and White Mclane Children's, Belton, Texas
  - Children's Memorial Hermann, Houston, Texas
  - Texas Children's Hospital - Main, Houston, Texas
  - Texas Children's Hosptial - West Campus, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Texas Children's Hospital The Woodlands, The Woodlands, Texas
  - Primary Children's Hospital - Lehi Campus, Lehi, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - WVU Children's Hospital, Morgantown, West Virginia
  - Children's Wisconsin, Milwaukee, Wisconsin
  - Children's Wisconsin - Fox Valley, Neenah, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Upon completion of the trial and after all planned analyses have been finalized, the research team will develop a de-identified public-use dataset. This dataset will include key variables necessary to replicate the primary analyses, along with accompanying documentation, such as data dictionaries and coding manuals. All personally identifiable information and protected health information will be removed prior to dataset release.